CLINICAL TRIAL: NCT02886793
Title: Cell Proliferation in Pulmonary Hypertension. FDG-PET Comparison Between Patients and Healthy Subjects
Acronym: PROCLAIM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joan Albert Barbera Mir (Other)
Responsible Party: Sponsor-Investigator, Joan Albert Barbera Mir, Dr, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-000347-14
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG (Experimental): all patients will undergo a PET scan and will receive 18F fludeoxyglucose
  Interventions: Drug: fludeoxyglucose

INTERVENTIONS:
Drug: fludeoxyglucose
  Other Names: FDG

SUMMARY:
Pulmonary arterial hypertension (PAH) and chronic thromboembolic pulmonary hypertension (CTEPH) are serious diseases with poor prognosis despite recent advances. Currently, pulmonary hypertension (PH) is considered a cell proliferative disorder, which has not been adequately characterized due to the lack of markers. A better understanding of the mechanisms that regulate this proliferative disorder will allow the identification of new therapeutic targets for HP.

The objective of the project is to identify cell proliferative processes in severe forms of PH. Patients with PAH (n=20), CTEPH (n=20) and healthy controls (n=20) will undergo characterization of microRNAs (miRNAs) contained within circulating microparticles (MPs) analysis and mitochondrial functionality and FDG-PET to compare cell metabolism in the lungs and the right ventricle between patients and controls.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PAH:

   * Hemodynamic diagnosis of precapillary pulmonary hypertension: PAPm ≥25 mmHg, PCWP ≤15 mmHg
   * Exclusion of group 2,3,4 or 5
2. Patients with CTEPH:

   * Hemodynamic diagnosis of precapillary pulmonary hypertension: PAPm ≥25 mmHg, PCWP ≤15 mmHg
   * Persistence of thrombotic perfusion defects on pulmonary scintigraphy or angioCT, after 3 months or more of correct anticoagulant therapy
3. Healthy subjects

   * No known disease or condition
   * Normal lung function, chest x-ray, EKG and blood chemistry and haematology

Exclusion Criteria:

* Severe comorbidity.
* Pulmonary, pleural or rib cage disease interfering with FDG-PET acquisition
* Malignancy with exception of basocellular carcinoma
* Current smoker or former smoker (last 10 years or more than 10-year-pack).
* Pregnant or lactating women Hyperglycemia (fasting above 200 mg/dL)
* Hypersensitivity to the product or its excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-06; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
FDG uptake in lung parenchyma | 1 hour

IPD SHARING:
Plan to Share IPD: No